CLINICAL TRIAL: NCT01703143
Title: A Pilot Study to Evaluate MR-guided Laser Ablation of Focal Lesions in Patients With Medically Refractory Partial Epilepsy
Brief Title: Pilot Study to Evaluate MR-guided Laser Ablation of Focal Lesions in Patients With Medically Refractory Partial Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, W. Richard Marsh, Principle Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007909
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser Ablation (Experimental): Laser ablation of focal lesions in patients with medically refractory partial epilepsy.
  Interventions: Procedure: Laser ablation

INTERVENTIONS:
Procedure: Laser ablation — Laser ablation of focal lesions in patients with medically refractory partial epilepsy.

SUMMARY:
To investigate whether MR-guided laser induced thermal therapy in patients diagnosed with focal lesional epilepsy using the Visualase Thermal Therapy System is both a feasible and safe minimally invasive technique for control of seizures in such patients.

DETAILED DESCRIPTION:
In this study, we propose to evaluate a novel, thermal therapy and feedback system (Visualase® Thermal Therapy System) as an alternative to surgical resection for the treatment of focal lesional epilepsy in patients that are considered high risk surgical candidates. This system includes the FDA-cleared Visualase Cooled Laser Applicator System (VCLAS), which allows delivery of laser energy while the patient is being imaged by an MRI unit. The Visualase® System works via real-time MR thermal imaging (MRTI) to provide information on the thermal dose delivered to the target, resulting in a more precise and controlled delivery which has heretofore not been possible with previous non-image guided laser technology. We hypothesize that the Visualase system can be used in patients refractory to medication therapy in a minimally invasive procedure to destroy epileptogenic focal lesions in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at entry to protocol.
* History of MRI lesional-related epilepsy for at least one year.
* Failure to respond to more than 2 anti-epileptic drugs at adequate dose and duration.
* Candidate for resective epilepsy surgery.
* Considered healthy enough to undergo surgery with general anesthesia.
* The patient has given written informed consent after the nature of the study and alternative treatment options have been explained.
* Must have 3 months of seizure frequency recorded prior to procedure.

Exclusion Criteria:

* Presence of any non-MRI compatible implanted electronic device.
* Presence of a metallic prosthetic or implant including artificial hips, knees, joints, or rods and screws.
* Active Major depression
* History of Suicide attempts
* History of Non-Epileptic Behavioral Spells

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The number of seizures recorded in seizure diary | Baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: W Marsh, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota